CLINICAL TRIAL: NCT01137890
Title: Effect of Zonisamide on Cocaine Reinforcement, Craving, and Relapse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R01DA027065 (NIH); R01DA027065 (NIH)
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Cocaine Dependence
Keywords: cocaine; addiction; drug dependence; anticonvulsant; zonisamide; drug self-administration; nicotine withdrawal; neurocognition
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive; Substance-Related Disorders | interventions — Zonisamide; Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonisamide (Experimental): Participants administered blind capsules containing either placebo or zonisamide.
  Interventions: Drug: Zonisamide; Drug: Cocaine Hydrochloride; Behavioral: Neurocognitive and Performance Battery; Behavioral: Smoking Assessments
- Placebo (Placebo Comparator): Participants administered only placebo capsules containing lactose.
  Interventions: Drug: Placebo; Drug: Cocaine Hydrochloride; Behavioral: Neurocognitive and Performance Battery; Behavioral: Smoking Assessments

INTERVENTIONS:
Drug: Zonisamide — Eight capsules administered daily in split doses at 22:00 and 09:00.
  Other Names: Zonegran,; CAS 68291-97-4,
  Arms: Zonisamide
Drug: Placebo — capsules administered in split doses at 22:00 and 09:00.
  Arms: Placebo
Drug: Cocaine Hydrochloride — Cocaine Challenge Sessions: Human laboratory sessions with administration of moderate doses of cocaine by the intravenous route under controlled conditions and cardiovascular monitoring.
  Other Names: CAS 50-36-2; methylbenzoylecgonine; benzoylmethylecgonine; C17H21NO4
Behavioral: Neurocognitive and Performance Battery — Participants will complete tests to assess their abilities and performances on a number of tasks given by a computer or other type of equipment.
Behavioral: Smoking Assessments — Participants answer questions about smoking and smoking behaviors are monitored.

SUMMARY:
This is a residential pilot trial to evaluate the pharmacodynamic interaction between zonisamide and cocaine, with the goal of evaluating zonisamide's potential for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
This is a residential pilot trial to evaluate the effect of zonisamide (ZNS) on cocaine reinforcement, craving and relapse. Cocaine addiction remains a major social and medical problem that imposes a significant burden on our society, as more than a half million cocaine dependent individuals are seeking treatment every year. Medications that act to antagonize the glutamate system and/or increase the GABA-system are new targets in the search towards effective cocaine treatment. ZNS is part of a new line of antiepileptic agents that act both as glutamate antagonists and to enhance the Gamma-AminoButyric acid (GABA) system. Topiramate, a similar agent, showed a positive signal in a pilot trial for cocaine dependence. ZNS has the advantages of a longer half-life requiring only once a day dosing and, being better tolerated, it requires a shorter induction phase and can be administered at higher doses. We hypothesize that ZNS in moderate to high doses will attenuate the central effect of cocaine and improve the neural perturbations resulting from cocaine use, thus decreasing cocaine craving. Healthy, adult cocaine dependent volunteers will be enrolled on our residential unit for 44 days for this double-blind within subject study. The pharmacodynamic interactions between ZNS and cocaine will be measured in cocaine self-administration procedure offering alternative reinforcers with monetary values. Cocaine reinforcing effect will be evaluated over a range of doses, and subjective and objective outcomes on mood and behavior will be collected. In addition, the effect of ZNS on ad-lib smoking will be studied on the days when no other procedure interferes with smoking behaviors. Neurocognitive and psychomotor effects of ZNS treatment will also be studied with an extensive test battery on the day of the week when no cocaine is administered. This study will explore the potential therapeutic effect of ZNS for the treatment of cocaine dependence while providing necessary safety assessments required for possible future outpatient clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 21 years old, not older than 45 years.
* Evidence of cocaine dependence.
* Not seeking treatment for cocaine abuse.
* Able and willing to be restricted to our unit for 6-7 weeks.
* Able to answer frequent questionnaires reliably and consistently.
* Smoker.

Exclusion Criteria:

* Allergy to Sulfonamide drugs (e.g. topiramate, zonisamide, sulfamethoxazole/trimethoprim).
* Diabetes, respiratory insufficiency, renal tubular acidosis or renal insufficiency, heart failure, liver insufficiency, chronic diarrhea, other chronic diseases predisposing to acidosis.
* Renal insufficiency defined as serum creatine > 1.30 mg/DL for males or > 1.03 mg/DL for females.
* History of nephrolithiasis, unexplained hematuria on screening urinalysis.
* History of head injury (with loss of consciousness longer than a few minutes).
* History of seizure, or use of antiepileptic medications.
* HIV positive individuals who meet AIDS by Centers for Disease Control (CDC) criteria or are on antiretroviral medications.
* BMI < 19 or BMI > 34.
* Total cholesterol > 240mg%.
* Serous psychiatric illness with psychosis, dementia.
* Glaucoma, family history of glaucoma, one-sided blindness.
* For female participants: being pregnant, lactating or not using an effective method of contraception.
* Physical dependence on any drug other than cocaine, nicotine, or caffeine.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Umbricht, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 14 | 5
Completed | 8 | 2
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (5.6) | 38.2 (4.1) | 38.7 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Questionnaire (VAQ) Score
Description: VAQ measures the change in effect after dose administration. Participants rate 6 items ("Any Drug Effect", "Rush", "Good Effects", "Bad Effects", "Liking", & "Desire for Cocaine") by pointing an arrow along a 100-point line anchored at either end with "none" (0) & "extremely" (100). Each participant's score is equal to the sum of all 6 ratings, & the mean of all participant's scores is reported across each condition. The VAQ is only administered to subjects in the zonisamide (Zon) condition (n=8). Repeated within-subject measures ANOVA performed to observe the main effects of Zon dose (0, 300, & 600mg) & cocaine dose (1, 20, & 40mg), & their interaction. All 8 subjects who received Zon completed both 300mg & 600mg doses. Assessments obtained on Week 1 (0mg Zon), Week 3 (300mg Zon), & Week 5 (600mg Zon), in which all 3 cocaine were co-administered at these times. Cocaine not administered (only Zon) during Weeks 2 & 4, thus no measures taken at these times
Time Frame: Weeks 1-5; mean of weeks 1, 3 and 5 reported
Population: Because we are interested in how co-administered of cocaine-Zon affects this measure, only Zon participants are included (n=8). Each participant receives varying doses of Zon (0, 300, 600mg) at weeks 1, 2-3, 4-5, respectively. After getting used to each Zon dose, they are co-administered all 3 cocaine doses (1, 20, 40mg) during Weeks 1, 3, and 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1mg-0mg: 1mg cocaine - 0mg zonisamide
  Both doses are expected to be inactive, thus this arm is viewed as Placebo
- 1mg-300mg: 1mg cocaine - 300mg zonisamide
- 1mg-600mg: 1mg cocaine - 600mg zonisamide
- 20mg-0mg: 20mg cocaine - 0mg zonisamide
- 20mg-300mg: 20mg cocaine - 300mg zonisamide
- 20mg-600mg: 20mg cocaine - 600mg zonisamide
- 40mg-0mg: 40mg cocaine - 0mg zonisamide
- 40mg-300mg: 40mg cocaine - 300mg zonisamide
- 40mg-600mg: 40mg cocaine - 600mg zonisamide
Arm/Group | 1mg-0mg | 1mg-300mg | 1mg-600mg | 20mg-0mg | 20mg-300mg | 20mg-600mg | 40mg-0mg | 40mg-300mg | 40mg-600mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 0.38 (0.74) | 3.75 (6.41) | 0.38 (0.74) | 40.63 (24.37) | 32.63 (14.78) | 30.00 (27.88) | 37.38 (21.84) | 29.75 (16.52) | 37.25 (25.47)
Statistical Analysis 1: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p < 0.01, ANOVA — p-value was calculated as less than 0.01. Note: this is not an attempt to indicate a threshold; F-value for main effect of Coc dose = 24.9 — F-value for main effect of Cocaine dose on VAQ score
Statistical Analysis 2: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.72, ANOVA; F-value for main effect of Zon dose = 0.34 — F-value for main effect of Zonisamide dose on VAQ score
Statistical Analysis 3: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.63, ANOVA; F-value for main effect of Coc x Zon = 0.66 — F-value for main effect of Cocaine x Zonisamide interaction on VAQ scores

2. Primary Outcome: Behavioral Choice Measures
Description: In each condition of cocaine-zonisamide dose, participants were asked to choose whether they would rather have a repeated cocaine dose (same dose as most recent administration) or cash of varying monetary value. The mean number of cocaine choices across each drug condition are reported. This measure only included participants in the zonisamide (Zon) condition (n=8), with each arm representing variation in co-administration of cocaine-Zon.
  Repeated within-subject measures ANOVA performed to observe the main effects of zonisamide dose (0, 300, and 600mg) and cocaine dose (1, 20, and 40mg), and their interaction. Only participants who received the active zonisamide medication (n=8) were included in this portion of the analysis.
  During self-administration sessions are every 15 min over 1hr45min period. Assessment on Weeks 1 (0mg Zon), 3 (300mg Zon), 5 (600mg Zon), in which varying cocaine doses co-administered. Cocaine not administered (only Zon) during Weeks 2 & 4
Time Frame: Weeks 1-5, mean of weeks 1, 3 and 5 reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of cocaine choices
Arm/Group | 1mg-0mg | 1mg-300mg | 1mg-600mg | 20mg-0mg | 20mg-300mg | 20mg-600mg | 40mg-0mg | 40mg-300mg | 40mg-600mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
number of cocaine choices | 0 (0) | 0 (0) | 0.25 (0.71) | 2 (2.67) | 2.38 (2.33) | 2.25 (2.05) | 3.5 (2.93) | 3 (2.2) | 3.38 (2.39)
Statistical Analysis 1: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p < 0.01, ANOVA — p-value was calculated as less than 0.01. Note: this is not an attempt to indicate a threshold; F-value for main effect of Coc dose = 9.91 — F-value for main effect of Cocaine dose on Behavioral Choice measure
Statistical Analysis 2: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.93, ANOVA; F-value for main effect of Zon dose = 0.07 — F-value for main effect of Zonisamide dose on Behavioral Choice measure
Statistical Analysis 3: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.92, ANOVA; F-value for main effect of Coc x Zon = 0.24 — F-value for main effect of Cocaine dose x Zonisamide dose interaction on Behavioral Choice measure

3. Primary Outcome: Cocaine Craving
Description: Cocaine craving measured by Cocaine Selectivity Severity Assessment (CSSA). The CSSA is a reliable and valid tool to measure cocaine withdrawal severity within a 24 hr period, and has been shown to predict treatment response in a treatment setting. Participants are asked to rate 18-items on a Likert scale 0-7, with composite scores ranging 0-126 and higher numbers indicative of more severe withdrawal. Mean scores on CSSA across 39-day time period are reported.
Time Frame: Day 1-39
Population: Includes all participants analyzed (n=12; 8 zonisamide, 4 placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 | Day 11 | Day 12 | Day 13 | Day 14 | Day 15 | Day 16 | Day 17 | Day 18 | Day 19 | Day 20 | Day 21 | Day 22 | Day 23 | Day 24 | Day 25 | Day 26 | Day 27 | Day 28 | Day 29 | Day 30 | Day 31 | Day 32 | Day 33 | Day 34 | Day 35 | Day 36 | Day 37 | Day 38 | Day 39
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
units on a scale
  Zonisamide | 27.88 (10.25) | 27.25 (15.29) | 25 (14.32) | 19.13 (8.63) | 17.88 (11.51) | 13.5 (8) | 12.75 (11.21) | 12.13 (9.85) | 13.75 (10.93) | 9.63 (8.99) | 11.75 (9.18) | 14.25 (11.41) | 12.38 (10.86) | 23.63 (31.01) | 26.75 (39.46) | 24.88 (39.41) | 25.38 (38.93) | 24.13 (39.47) | 25.13 (39.67) | 12.75 (12.74) | 25.5 (29.82) | 15.25 (14.27) | 16.88 (12.05) | 13.88 (13.07) | 8.25 (9.41) | 10.25 (11) | 10.75 (10.17) | 7.63 (9.78) | 7.63 (10.82) | 6.57 (10.13) | 9.50 (9.09) | 11.25 (12.90) | 8.5 (10.43) | 13.5 (11.49) | 21.38 (17.74) | 8.13 (11.76) | 23.25 (35.25) | 8.25 (11.99) | 19.25 (27.22)
  Placebo | 42.75 (11) | 41 (20.54) | 30.25 (23.49) | 28.25 (15.73) | 28.25 (14.57) | 26.5 (9.32) | 29.5 (6.35) | 27.25 (11.87) | 28.5 (13.82) | 19 (9.93) | 25.33 (5.85) | 25.25 (15.6) | 22.75 (5.12) | 22.75 (9.74) | 24.75 (14.5) | 19.25 (5.25) | 24.00 (11.53) | 22.5 (12.36) | 24.5 (15.86) | 26 (15.490) | 25.5 (18.21) | 23 (15.09) | 18 (9.17) | 19 (0) | 15.5 (0.70) | 16. (2.83) | 14.5 (2.12) | 16.5 (3.53) | 24 (0) | 16.5 (0.71) | 16.5 (0.71) | 19.5 (4.95) | 18. (2.83) | 17. (1.41) | 19. (7.07) | 16 (0) | 19 (4.24) | 20 (4.24) | 16.5 (2.12)
Statistical Analysis 1: Comparison: Day 1 vs Day 2 vs Day 3 vs Day 4 vs Day 5 vs Day 6 vs Day 7 vs Day 8 vs Day 9 vs Day 10 vs Day 11 vs Day 12 vs Day 13 vs Day 14 vs Day 15 vs Day 16 vs Day 17 vs Day 18 vs Day 19 vs Day 20 vs Day 21 vs Day 22 vs Day 23 vs Day 24 vs Day 25 vs Day 26 vs Day 27 vs Day 28 vs Day 29 vs Day 30 vs Day 31 vs Day 32 vs Day 33 vs Day 34 vs Day 35 vs Day 36 vs Day 37 vs Day 38 vs Day 39; Test type: Superiority; p = 0.16, t-test, 2 sided — Group (Zonisamide vs Placebo); t-value for main effect of Group = 1.51
Statistical Analysis 2: Comparison: Day 1 vs Day 2 vs Day 3 vs Day 4 vs Day 5 vs Day 6 vs Day 7 vs Day 8 vs Day 9 vs Day 10 vs Day 11 vs Day 12 vs Day 13 vs Day 14 vs Day 15 vs Day 16 vs Day 17 vs Day 18 vs Day 19 vs Day 20 vs Day 21 vs Day 22 vs Day 23 vs Day 24 vs Day 25 vs Day 26 vs Day 27 vs Day 28 vs Day 29 vs Day 30 vs Day 31 vs Day 32 vs Day 33 vs Day 34 vs Day 35 vs Day 36 vs Day 37 vs Day 38 vs Day 39; Test type: Superiority — Day (Day 1-39); p = 0.0015, t-test, 2 sided; t-value for main effect of Day = -3.2
Statistical Analysis 3: Comparison: Day 1 vs Day 2 vs Day 3 vs Day 4 vs Day 5 vs Day 6 vs Day 7 vs Day 8 vs Day 9 vs Day 10 vs Day 11 vs Day 12 vs Day 13 vs Day 14 vs Day 15 vs Day 16 vs Day 17 vs Day 18 vs Day 19 vs Day 20 vs Day 21 vs Day 22 vs Day 23 vs Day 24 vs Day 25 vs Day 26 vs Day 27 vs Day 28 vs Day 29 vs Day 30 vs Day 31 vs Day 32 vs Day 33 vs Day 34 vs Day 35 vs Day 36 vs Day 37 vs Day 38 vs Day 39; Test type: Superiority — Group*Day interaction; p = 0.10, t-test, 2 sided; t value for Group x Day interaction = -1.63

4. Secondary Outcome: Drug Value Questionnaire
Description: Street Value of Sampled Dose. After co-administration of cocaine-zonisamide, participants were asked to hypothetically estimate the value of the drug they received, if they were to purchase it on the street. The mean value (dollars) across all drug conditions is reported here.
  Repeated within-subject measures ANOVA performed to observe the main effects of zonisamide dose (0, 300, and 600mg) and cocaine dose (0, 20, and 40mg), and their interaction. Only participants who received the active zonisamide medication (n=8) were included in this portion of the analysis. Additionally, all 8 subjects who received zonisamide completed both 300mg and 600mg doses.
  Within-subject repeated interval during self-administration sessions. Cocaine not administered (only Zon) during Weeks 2 & 4, thus no measures taken at these times
Time Frame: Weeks 1-5; mean of weeks 1, 3 and 5 reported
Population: Because we are interested in how co-administration cocaine-zon affects this measure, only zon participants are included (n=8). Each participant receives varying doses of zon (0, 300, 600mg) at weeks 1, 2-3, 4-5, respectively. After getting used to each zon dose, they are co-administered all 3 cocaine doses (1, 20, 40mg) during Weeks 1, 3, and 5
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | 1mg-0mg | 1mg-300mg | 1mg-600mg | 20mg-0mg | 20mg-300mg | 20mg-600mg | 40mg-0mg | 40mg-300mg | 40mg-600mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
dollars | 0 (0) | 0 (0) | 0 (0) | 9.29 (7.32) | 8.50 (5.81) | 7.63 (3.54) | 16 (14.96) | 18.13 (18.31) | 9.5 (8.57)
Statistical Analysis 1: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p < 0.01, ANOVA — p-value was calculated as less than 0.01. Note: this is not an attempt to indicate a threshold; F-value for main effect of Coc dose = 21.1 — F-value for main effect of Cocaine dose
Statistical Analysis 2: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.48, ANOVA; F-value for main effect of Zon dose = 0.77 — F-value for main effect of Zonisamide dose
Statistical Analysis 3: Comparison: 1mg-0mg vs 1mg-300mg vs 1mg-600mg vs 20mg-0mg vs 20mg-300mg vs 20mg-600mg vs 40mg-0mg vs 40mg-300mg vs 40mg-600mg; Test type: Superiority; p = 0.46, ANOVA; F-value for the main effect of Zon x Coc = 0.93 — F-value for main effect of Zonisamide x Cocaine interaction on drug value (i.e., street value) measurement

ADVERSE EVENTS:
Time Frame: 39 days
Description: Reported adverse events (AEs) include participants who were randomized into the study's conditions (zonisamide/placebo), and of which were rated as being either possibly, probably, or definitely related to the study.
  Although 19 participants were randomized, 9 did not complete. However, 2 of these provided sufficient data to be included in analyses. Thus, the possibility of study related AEs could only occur in 12 subjects (8 zonisamide, 4 placebo). This is the case for serious AEs, too.
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=8) | Placebo (N=4)
Allergic Rhinitis (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 6 (9) | 2 (4)
Inguinal Hernia (General disorders) | 1 (1) | 0 (0)
Skin Rash (General disorders) | 0 (0) | 1 (1)
Creatinine Elevation (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Appetite Decreased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hepatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver function abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth Disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chemistry Abnormal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain lower extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tingling sensation in extremity (Nervous system disorders) | 1 (2) | 0 (0)
Agitation (Nervous system disorders) | 0 (0) | 2 (2)
Dream abnormal (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Jittery (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (General disorders) | 1 (1) | 1 (1)
Rhinitis (General disorders) | 0 (0) | 1 (1)
Athlete's foot (General disorders) | 1 (1) | 0 (0)
Tinnitus (Eye disorders) | 1 (1) | 0 (0)
Urethritis (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No